CLINICAL TRIAL: NCT02768311
Title: Comparative Evaluation of Post Endodontic Pain Following Root Canal Treatment With Two Rotary System: Neolix & Waveone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7354
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-04

CONDITIONS: Pain, Postoperative Pain Pathologic Processes Postoperative Complications Signs and Symptoms
Keywords: Instrumentation Post-operative pain Root canal preparation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- neolix rotary system (continuous rotation system) (Experimental): Procedure: neolix rotary system post-treatment pain after using neolix rotary system
  Interventions: Procedure: neolix rotary system (continuous rotation system)
- waveone rotary system (reciprocating system) (Experimental): Procedure: waveone rotary system post-treatment pain after using waveone rotary system
  Interventions: Procedure: waveone rotary system (reciprocating system)
- hand files k-files (Experimental): Procedure: hand files post-treatment pain after using hand files
  Interventions: Procedure: hand files k-files

INTERVENTIONS:
Procedure: neolix rotary system (continuous rotation system) — Procedure: neolix rotary system
  Arms: neolix rotary system (continuous rotation system)
Procedure: waveone rotary system (reciprocating system) — Procedure: waveone rotary system
  Arms: waveone rotary system (reciprocating system)
Procedure: hand files k-files — Procedure: hand files k-files
  Arms: hand files k-files

SUMMARY:
Today, dentists tend to use rotary systems. Despite the increasing diversity of these systems as well as a few studies on the prevalence of pain after root canal treatment by rotary systems, And in particular, comparing the amount of pain after treatment, between systems RECIPROCAL AND FULL ROTATION single-file, the aim of this study was to evaluate the effect of applying canal preparation by the system, Neolix and WaveOne, on the prevalence of pain after endodontic treatments.

DETAILED DESCRIPTION:
Many studies of pain after root canal treatment experience were taken into consideration.

Pain after endodontic treatment is still one of the major problems of patients. The prevalence that widely studied as 6/10% to 9.82% have been reported.

One of the important strategies in endodontic treatment, prevention and control of pain after treatment. This multi-factorial disorder resulting in a complex process occurs, which affects the patient's intrinsic factors, the tooth and the dentist's skill.

Mechanical factors include channel instrumentation techniques, over instrumentation or filling material extrusion channels associated with the presence of pain after treatment were considered.

Apical extrusion of infected debris during instrumentation channel can create or exacerbate inflammatory process. Channel shaping the apical debris extrusion process can increase even if the preparation is limited to the channel. Leaving debris in both methods of preparation, either manually with stainless steel files and rotary technique with nickel titanium files happen.

The use of rotary technique among dentists has increased. developing of NITI files and rotary instrumentation system, reduce apical extrusion of debris, so can be expected to reduce the incidence of inflammation and pain after treatment, achieved by these means.

Recent studies have shown that reciprocal shaping techniques, compared with full-rotation techniques, significantly increased the amount of debris extruded from the apical region of the root are causing increasing pain after treatment.

Two rotary system available on the market are:

1) Neolix (france Neolix SAS) recently introduced the file NITI, single file, with full rotation movements, with square and rectangular cross-section, with a non-uniform shape along the blade, tip sizes, 25 and Tipper 0 / 08, and a system, Wave one, (DENTSPLY Maillefer), which is a file NITI, Single file and Single use, and the reciprocation movements, and cross-Convex triangular Modified and in three sizes: small, primary (tip size 25 and Tipper 0/08), large is contained, which according to the size of the canal, one of them is selected.

In a study by Ana Arias et al., Patients in the experimental group by the Rotary Files roots were treated and patients in control group were treated by the step-back technique, the results showed that more patients in the control group, experienced pain after root canal therapy. While the duration of the pain in the control group comparison to the experimental group, less has been reported.

In a study by Aqrabawi, teeth with vital pulp were divided into two groups. Root canal therapy in the first group, was done by manual file, and the second group, by Protaper rotary files were performed.

And no significant difference in pain after root canal treatment has not been detected.

Gambarini was shown in the study, patients treated by waveone system they have done, significantly more pain after treatment compared to TF and TF adaptive experienced.

Today, dentists tend to use rotary systems. Despite the increasing diversity of these systems as well as a few studies on the prevalence of pain after root canal treatment by rotary systems, And in particular, comparing the amount of pain after treatment, between systems RECIPROCAL AND FULL ROTATION single-file, the aim of this study was to evaluate the effect of applying canal preparation by the system, Neolix and WaveOne, on the prevalence of pain after endodontic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-50 years,
* the systemically healthy,
* first or second molar teeth require root canal therapy,
* irreversible Pulpitis signed without the apical,
* root canal curvature of less than 25 degrees, according to Schneider techniques.

Exclusion Criteria:

* Root canal treatment,
* history of medication (antibiotics, NSAID, opiates) of the patient 12 hours before treatment,
* pregnancy,
* complex anatomy,
* channels blocked in the x-ray plate,
* internal and external resorption,
* open apex teeth,
* periodontal disease,
* inflammation and abscesses,
* sinus tract,
* presence of radiographic lesions,
* tooth sensitivity to percussion,
* absence of occlusal contact.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Information regarding post-operation pain is gathered via a patient using questionnaire and is measured via the visual analogue scale | 12 month

IPD SHARING:
Plan to Share IPD: Yes